CLINICAL TRIAL: NCT05632354
Title: An Open-label Extension Study to Evaluate the Long-term Safety of GBT021601 Administered to Participants With Sickle Cell Disease Who Have Participated in a GBT021601 Clinical Trial
Brief Title: GBT021601-022: A Study of GBT021601 in Participants With Sickle Cell Disease (SCD)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study terminated as data obtained from this non-placebo-controlled trial may not be informative for the interpretation of the benefits and risks of osivelotor
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBT021601-022; C5351005 (Other: Alias Study Number)
Record Dates: First submitted 2022-11-01; First posted 2022-11-30 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Osivelotor
  Interventions: Drug: Osivelotor

INTERVENTIONS:
Drug: Osivelotor — Osivelotor

SUMMARY:
An Open-label Extension Study of GBT021601 in Participants with Sickle Cell Disease

DETAILED DESCRIPTION:
An Open-label Extension Study to Evaluate the Long-term Safety and Efficacy of GBT021601 Administered to Participants with Sickle Cell Disease Who Have Participated in a GBT021601 Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 6 months or older with SCD who participated and received study drug or placebo in a previous osivelotor clinical study and completed the end of treatment visit.

   Note: Participants who discontinued study drug in the originating study due to an TEAE, but who remained on study, may be eligible for treatment in this study provided the TEAE does not pose a risk for treatment with osivelotor.
2. Females of childbearing potential are required to have a negative urine pregnancy test prior to dosing on Day 1.

   Note: Females who become of childbearing potential during the study must be willing to have negative urine pregnancy tests to remain in the study.
3. If sexually active, females of childbearing potential must consistently use highly effective methods of contraception consistently throughout the study and for at least 120 days after the last dose of study drug. If sexually active, male participants must use barrier methods of contraception until 84 days after the last dose of study drug. Male participants are eligible to participate if they agree to the following requirements during the study intervention period and for 84 days after the last dose of study intervention:

   * Refrain from donating sperm PLUS either
   * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle OR
   * Must agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person
4. Participant has provided written informed consent/assent. For underage participants, both the consent of the participant's legal representative or legal guardian and the participant's assent (where applicable) must be obtained based on local requirements.

Exclusion Criteria:

* Participant withdrew consent or was noncompliant from the originating osivelotor clinical study
* Current or recent use of voxelotor. Recent use is defined as within 10 days prior to Day 1
* Current or recent use of crizanlizumab. Recent use is defined as within 90 days prior to Day 1
* Participant has any medical, psychological, safety, or behavioral conditions that, in the opinion of the Investigator, may confound safety interpretation, interfere with compliance, or preclude informed consent
* Has received an investigational drug (including investigational vaccines) within 5 times the elimination half-life (if known) or within 30 days (if the elimination half-life- is unknown) prior to study drug administration or is concurrently enrolled in any research judged not to be scientifically or medically compatible with this study

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | From time of enrollment through end of treatment up to 5 years
  Treatment-Emergent Adverse Events
Changes in laboratory assessments | From time of enrollment through end of treatment up to 5 years
  Safety laboratory data observed values and change from baseline
Changes in Vital signs | From time of enrollment through end of treatment up to 5 years
  Vital signs observed values and change from baseline

SECONDARY OUTCOMES:
Annualized rate of VOC | From time of enrollment through end of treatment up to 5 years
  Annualized rate of vaso-occlusive crisis will be calculated
Incidence of SCD-related SAEs | From time of enrollment through end of treatment up to 5 years
  Incidence of Sickle Cell Disease-related serious adverse events
Change from baseline in hematological laboratory parameters | From time of enrollment through end of treatment up to 5 years
  Hematological laboratory parameters will include hemoglobin, reticulocytes, lactate dehydrogenase, and unconjugated bilirubin.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (5):
  - Our Lady of the Lake Hospital, Inc., Baton Rouge, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - University of Texas Health Science Center, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
- Nigeria (3):
  - University College Hospital Ibadan, Ibadan, Oyo/ibadan North
  - Aminu kano Teaching Hospital, Kano
  - Lagos University Teaching Hospital, Lagos

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT021601-022